CLINICAL TRIAL: NCT00172679
Title: Effects of Tai Chi Exercise on Innate and Adaptive Immune Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361701225
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2004-12

CONDITIONS: Healthy
Keywords: Tai Chi; NK Cells; T lymphocytes; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Tai Chi is a traditional Chinese martial art that has been practiced for many centuries. Improvements in cardiorespiratory function, balance, muscular strength, flexibility in older subjects; preventing falls in the frail elderly; stress reduction, and mood state with Tai Chi practices have been well established. A potential immune response effect of Tai Chi practice is a frequent claim; however, this is an under-researched area. Therefore, in this study, the researchers will examine the effects of Tai Chi on innate and adaptive immune function.

DETAILED DESCRIPTION:
Tai Chi, a traditional Chinese martial art that has been practiced for many centuries, has only recently gained the interest of researchers in Western countries as an alternative form of exercise. Tai Chi combines deep diaphragmatic breathing and relaxation with many fundamental postures that flow imperceptibly and smoothly from one to the other through slow, gentle, and graceful movements. Based on the maximum oxygen consumption (VO2max) measured during the practice, Tai Chi is characterized as a low- to moderate-intensity form of exercise. Tai Chi has been applied as a rehabilitation program in patients with heart failure, hypertension, acute myocardial infarction, arthritis, and multiple sclerosis. Improvements in cardiorespiratory function, balance, muscular strength, flexibility in older subjects; preventing falls in the frail elderly; stress reduction, and mood state with Tai Chi practices have been well established. A potential immune response effect of Tai Chi practice is a frequent claim; however, this is an under-researched area. A nonrandomized controlled study of 60 elderly subjects found that the total number of circulating T cells were significantly higher in the Tai Chi group (who regularly practiced Tai Chi for 4 or more years) than in the untrained group. Irwin et al. demonstrated that older adults with no previous Tai Chi experience after practicing for 15 wks (1-3 times/wk), a nearly 50% increase in varicella zoster virus specific, cell-mediated immunity was found. Thus in this proposed study, we will examine the effects of regular Tai Chi practitioners on innate and adaptive immune function.

ELIGIBILITY:
Inclusion Criteria:

* Has been practicing Tai Chi Chuan (TCC) for at least 3 days a week for at least 12 months.

Exclusion Criteria:

* Any chronic systemic diseases (e.g., coronary artery disease [CAD])
* Has cognitive impairments.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, Ph.D., Principal Investigator — National Taiwan University, College of Medicine
Locations (2):
- Taiwan (2):
  - School & Graduate Institute of Physical Therapy, College of Medicine, NTU, Taipei, Taipei
  - National Taiwan University Hospital, Taipei